CLINICAL TRIAL: NCT06990035
Title: Implementazione di un Intervento Multiplo Per Promuovere Stili di Vita Sani in Pazienti Con Depressione: Uno Studio Clinico Controllato e Randomizzato
Brief Title: Implementation of a Multiple Intervention to Promote Healthy Lifestyles in Patients With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5M-2022-23685026
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major depressive disorder; Physical activity; Mediterranean Diet; Microbiome
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Mediterranean diet lessons program
  Interventions: Behavioral: Mediterranean diet lessons program
- Experimental Group (Experimental): Physical activity program
  Interventions: Behavioral: Mediterranean diet lessons program; Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Mediterranean diet lessons program — Participants will attend five one-hour lessons delivered by qualified professionals to learn about foods that have a positive impact on cognitive function and how to incorporate them into their dietary regimen.
Behavioral: Physical activity — Participants will undergo a 12-week physical exercise program guided by specified personal trainers.
  Arms: Experimental Group

SUMMARY:
This clinical trial aims to investigate whether an integrative approach combining education on the Mediterranean diet and physical activity (PA) can significantly reduce depressive symptomatology in individuals with major depressive disorder. The study will evaluate changes in depressive symptoms and assess biological modulations, including alterations in the gut microbiota and inflammatory markers, resulting from the PA intervention.

Participants will be randomized into two arms: the active control group will attend a series of lessons focused on the Mediterranean diet, while the experimental group will participate in the same dietary lessons combined with a structured PA program of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of depression (DSM-5 criteria, American Psychiatric Association 2013).
* Depressive symptoms assessed using MADR, BDI, or ZDR scales.
* Ability to provide written informed consent.
* Self-reported moderate-intensity leisure physical activity of less than 150 minutes per week.

Exclusion Criteria:

* Patients with severe psychopathology.
* Medical contraindications to physical activity.
* Orthopedic problems or other conditions limiting physical fitness assessment or currently pregnant.
* Patients who underwent antibiotic/anti-inflammatory treatments in the last 3 months
* Active gastrointestinal diseases
* Autoimmune and/or chronic inflammatory disorders

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
MADR Scale for Depression | Baseline (day 1); Week 6 (up to 6 weeks, mid-treatment); Week 12 (up to 12 weeks, end of treatment).
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-administered scale designed to assess the severity of depressive symptoms. It consists of 10 items, each rated on a scale from 0 to 6, yielding a total score ranging from 0 to 60. Higher scores indicate greater severity of depression, meaning a worse clinical outcome.
Beck Depression Inventory - II | Baseline (day 1); Week 6 (up to 6 weeks, mid-treatment); Week 12 (up to 12 weeks, end of treatment).
  The Beck Depression Inventory (BDI) is a self-report questionnaire used to assess the presence and severity of depressive symptoms. It comprises 21 items, each rated on a scale from 0 to 3, resulting in a total score ranging from 0 to 63. Higher scores reflect more severe depressive symptoms, indicating a worse clinical outcome.
Zung Self-Rating Depression Scale | Baseline (day 1); Week 6 (up to 6 weeks, mid-treatment); Week 12 (up to 12 weeks, end of treatment).
  The Zung Self-Rating Depression Scale (ZRS) is a self-administered questionnaire designed to assess the level of depressive symptoms in individuals. It consists of 20 items, each rated on a scale from 1 to 4, based on how often symptoms are experienced. The raw total score ranges from 20 to 80, which is often converted to an index score (ranging from 25 to 100) by multiplying the raw score by 1.25. Higher scores indicate more severe depression
Personal and Social Performance Scale | Baseline (day 1); Week 6 (up to 6 weeks, mid-treatment); Week 12 (up to 12 weeks, end of treatment).
  The Personal and Social Performance Scale (PSP) is a clinician-rated instrument used to assess personal and social functioning in individuals with mental disorders. The total score ranges from 1 to 100, with higher scores indicating better functioning and a more favorable clinical outcome.
World Health Organization Quality of Life - Bref | Baseline (day 1); Week 6 (up to 6 weeks, mid-treatment); Week 12 (up to 12 weeks, end of treatment).
  The WHOQOL-BREF is a self-report questionnaire developed by the WHO to assess quality of life across multiple domains. It contains 26 items rated on a 5-point Likert scale. Higher scores indicate a better quality of life, reflecting a more favorable outcome.

SECONDARY OUTCOMES:
Immunitary-related factors levels | Baseline (day 1); Week 12 (up to 12 weeks, end of treatment).
  Plasma/serum levels of cytokines
Gut Microbiome Composition | Baseline (day 1); Week 12 (up to 12 weeks, end of treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro San Giovanni fi Dio Fatebenefratelli, Brescia, Italy